CLINICAL TRIAL: NCT06585007
Title: Metastasis-directed Therapy in Oligoprogressive Castration-refractory Prostate Cancer: a Randomized Phase 3 Trial
Brief Title: Metastasis-directed Therapy in Oligoprogressive Castration-refractory Prostate Cancer
Acronym: MEDCARE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S67130; 2022-502254-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-22; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-04

CONDITIONS: Castration-resistant Prostate Cancer; Oligoprogressive
MeSH Terms: interventions — Radiotherapy; Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care therapy (No Intervention): The standard of care can consist of surveillance (which means the continuation of the ongoing systemic treatment without any change) or initiation of NEST. The decision which option is considered must be decided at the multidisciplinary urologic oncology meeting (obligatory). MDT is not allowed in this arm. Options for NEST in this trial are abiraterone acetate, enzalutamide, apalutamide, darolutamide, olaparib, talazoparib, niraparib, cabazitaxel and docetaxel, radium-223, luthetium-177-PSMA.
- Progression-directed therapy (Experimental): PDT (metastasectomy or SBRT) while continuing current systemic therapy: androgen-deprivation (ADT) alone, or ADT in combination with abiraterone acetate, enzalutamide, apalutamide and patients who had received docetaxel in the past. Patients under current treatment with docetaxel are not allowed, because the hypothesized interaction between docetaxel and radiotherapy concerning toxicity. In case of oligoprogression after PDT, repeated PDT to the new lesions is mandatory.
  Interventions: Radiation: Radiotherapy; Procedure: metastasectomy

INTERVENTIONS:
Radiation: Radiotherapy — Progression-directed therapy (stereotactic body radiation therapy)
  Arms: Progression-directed therapy
Procedure: metastasectomy — Progression-directed therapy (metastasectomy)
  Arms: Progression-directed therapy

SUMMARY:
Evaluation of the impact of metastasis-directed therapy in patients with castration-refractory prostate cancer and a maximum of 5 progressive lesions.

DETAILED DESCRIPTION:
MEDCARE phase 3 trial is approved by the central Ethics committee. It is a multicentric, randomized, prospective, open-label, two-arm, phase III trial. The aim is to evaluate the impact of progression-directed therapy (PDT) in patients presenting with oligoprogressive mCRPC on overall survival (OS). The study will employ a 1:1 randomization between arm A and arm B. Patients will be stratified according to number of metastases (1 versus > 1), initial localization (local recurrence, N or M1a vs. M1b or M1c) and systemic therapy (patient type 1 vs. type 2, see below) (Fig 1). Randomization will be carried out after approval in the multidisciplinary tumour board were the standard-of-care treatment and kind of PDT (metastasectomy or SBRT) will be decided before randomization.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this Trial must meet all the following criteria:

* Written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
* Acinar adenocarcinoma (inclusive neuro-endocrine dedifferentiation).
* Oligoprogressive disease on conventional imagine within a maximum of 6 weeks prior to randomisation defined as: a maximum of 3 extracranial progressive lesions (pre-existing lesions, the development of new lesions, or both) in any organ. Nodal (N1) disease should be measured in the short axis. Nodes more than 1.5 cm in the short axis are considered pathologic and measurable. Oligoprogression on bone scan is defined as the occurrence of maximal 3 new and/or progressive lesions. In case of not unambiguously, additional imaging such as diagnostic magnetic resonance imaging (MRI) or dedicated CT-scan should be performed. Visceral disease reported separately (lung, liver, adrenal, or CNS) and is considered measurable if an individual lesions is more than 1 cm longest dimension.

In case of locally persistent/recurrent disease, a diagnostic MRI of the prostate (bed) and/or biopsy of the site is recommended. There are two different mCRPC patient groups who are eligible for inclusion in the trial:

1. Patients with oligoprogressive disease with pADT only as ongoing treatment (Type 1).
2. Patients with oligoprogressive disease with pADT +/- second line systemic therapy. This is both the combination of pADT + ARTA as ongoing treatment or patients who had received docetaxel in the past (Type 2).

   * Castration-refractory disease, defined as testosterone level < 50 ng/dL.
   * Prior treatment of the primary tumor by radiotherapy or surgery. If the primary tumor has not been treated previously, this treatment is obligatory within the trial.
   * WHO performance 0-2
   * Age >= 18 years old
   * Absence of psychological, sociological, or geographical condition potentially hampering compliance with study protocol.
   * Patients must be presented at the multidisciplinary board meeting and the inclusion in the trial needs approval by this board.

Exclusion Criteria:

* Ductal adenocarcinoma and small-cell prostate cancer.
* Serum testosterone level > 50 ng/ml.
* Presence of poly-progressive disease, defined as more than 3 progressive lesions on conventional imaging or nodal and/or metastatic lesions on conventional imaging
* Active malignancy other than prostate cancer that could potentially interfere with the interpretation of this trial.
* Previous treatments (RT, surgery) or comorbidities rendering new treatment with SBRT impossible.
* Spinal bone lesion that is highly symptomatic, neurologically threatening or at risk of fracture.
* Patients already treated with radionuclides, cabazitaxel or PARP-inhibitors in the past.
* Patients with progressive disease while receiving docetaxel.
* Not able to understand the treatment protocol or sign informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2029-01-20 (Estimated); Study Completion 2029-01-20 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | will be calculated from the day of randomisation until death from any cause, wichever came first, assessed up to 5 years.
  Overall Survival

SECONDARY OUTCOMES:
Quality of life scoring EORTC QLQ-C30 | Assessments are planned at baseline and during follow-up consultation at month 1, month 3, month 6, month 12 and month 24
  Quality of life scoring using the EORTC QLQ-C30
Quality of life scoring EORTC QLQ-PR25 | Assessments are planned at baseline and during follow-up consultation at month 1, month 3, month 6, month 12 and month 24
  Quality of life scoring using the EORTC QLQ-PR25
Quality of life scoring EQ-5D-5L | Assessments are planned at baseline and during follow-up consultation at month 1, month 3, month 6, month 12 and month 24
  Quality of life scoring using the EQ-5D-5L.
Cancer Specific Survival | will be calculated from the day of randomisation until prostate cancer death, assessed up to 5 years.
  Cancer Specific Survival
Radiographic progression free survival | will be calculated from the day of randomisation until the first day of progression (local, nodal or metastatic). Imaging is performed every 6 months during follow-up or at any time in case of PSA progression or symptoms, assessed up to 5 years.
  Radiographic progression free survival
Progression-directed therapy induced acute or late toxicity scoring | Toxicity will be scored every follow-up visit, assessed up to 5 years after progression-directed therapy.
  Acute and late toxicity as a result of radiotherapy will be scored using the Common Toxicity Criteria Version 5.0 and metastasectomy related toxicity will be scored using Clavien Dindo scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT06585007/ICF_000.pdf